CLINICAL TRIAL: NCT06828731
Title: Sodium-glucose Transporter 2 Inhibitor Use in Pre-diabetes: Initial Evaluation in Veterans
Brief Title: Evaluation of Empagliflozin vs Standard Care in Veterans With Prediabetes
Acronym: PREVNT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charles George VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Beth Greck, Principal Investigator, Charles George VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00001926S01; VISN6CDA2024 (Other: Veterans Integrated Service Network 6 (Mid-Atlantic) Career Development Award)
Record Dates: First submitted 2024-11-21; First posted 2025-02-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (Active Comparator): Participants in this arm will receive lifestyle education to manage pre-diabetes as well as the monitoring of HbA1c, kidney function, weight, and blood pressure.
  Interventions: Other: Lifestyle education
- Standard Care plus empagliflozin (Experimental): Participants in this arm will receive lifestyle education to manage pre-diabetes as well as the monitoring of HbA1c, kidney function, weight, and blood pressure. They will also receive empagliflozin 10mg daily.
  Interventions: Drug: Empagliflozin 10mg daily; Other: Lifestyle education

INTERVENTIONS:
Drug: Empagliflozin 10mg daily — This intervention will assess recruitment and retention (feasibility trial).
  Arms: Standard Care plus empagliflozin
Other: Lifestyle education — This intervention is considered standard care for prediabetes.

SUMMARY:
Prediabetes effects 96 million people 18 years of age or older. It is important to identify treatment options to slow or prevent progression to diabetes. It is also critical to assess the potential of medications like sodium glucose transporter 2 inhibitors to reduce the risk of cardiovascular events and kidney complications, both common and costly complications of diabetes. This is a 12-week, open-label pilot feasibility study assessing the use of empagliflozin in prediabetes.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of prediabetes defined by HbA1c >5.7% and <6.5% or fasting glucose 100-125 mg/dL with documentation of diagnosis (ICD-10 code) within electronic health record at time of enrollment

* Age 35 to 60 years at time of enrollment
* Able to read and speak English

Exclusion Criteria:

* Diagnosis of diabetes (type 2 or type 1)
* Contraindication to SGLT2i medication per medication labeling, prior adverse reaction to SGLT2i medication, or received SGLT2i medication within the 6 months prior to enrollment
* Currently prescribed an antihyperglycemic agent approved for treatment of type 2 diabetes or taking any FDA-approved weight loss agent or over-the-counter supplement promoted for weight loss
* Veterans unable to complete informed consent process (Veterans with impaired decision-making ability or who require use of a legally authorized representative)
* Women who are pregnant or may become pregnant
* Veterans with neurogenic bladder, indwelling catheter, or urinary tract infection within the previous 12 months requiring hospitalization or emergency department visit

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Recruitment | 12 weeks
  Number of participants screened during study period Number of participants randomized during study period Number of participants enrolled during study period
Retention | 12 weeks
  Number of participants enrolled who complete the study Number of participants enrolled who do not complete the study and reason for not completing the study

SECONDARY OUTCOMES:
HbA1c (%) | 12 weeks
  HbA1c measured at baseline (visit 1) and 12 weeks (visit 3) will be reported as aggregate data for change from baseline to visit 3 for control group and exposure group.
Renal function (ml/min) | Every visit (baseline (T), T+2-4 weeks, T+12 weeks)
  estimated GFR (eGFR) (ml/min) will be collected at each study visit and reported as aggregate data for change from baseline to visit 2 and visit 3 for control group and exposure group.
Weight (kg) | Every visit (baseline (T), T+2-4 weeks, T+12 weeks)
  Weight (kg) will be collected at each study visit and reported as aggregate data for change from baseline to visit 2 and visit 3 for control group and exposure group.
Blood pressure (mmHg) | Every visit (baseline (T), T+2-4 weeks, T+12 weeks)
  Average of 2 sitting blood pressure measurements (mmHg) will be collected at each study visit and reported as aggregate data for change from baseline to visit 2 and visit 3 for control group and exposure group.
Adverse Events | 12 weeks
  Total number of adverse events occurring among enrolled participants in each group as well as type of adverse event. At conclusion of study will report percent of adverse events reported with each group, i.e. number of participants in control group reporting adverse event/total number of participants enrolled in control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Charles George VA Medical Center, Asheville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT06828731/ICF_000.pdf